CLINICAL TRIAL: NCT04147663
Title: Epidemiology of Suspected Epileptic Seizures
Acronym: EPI-lepsie
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Collaborators: RESCUe - RESeau Cardiologie Urgence / RESUVal - RESeau des Urgences de la vallée du Rhône (Other)
Responsible Party: Sponsor
Other Study IDs: EPILEPSIE2019
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Epilepsy
Keywords: emergency; epileptic seizure; epilepsy; neurology
MeSH Terms: conditions — Epilepsy; Emergencies; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: describe the management of the adult population suffering from suspected seizure by the emergency structures — For 3 consecutive days, all patients with suspected epileptic seizures (assessed by the Emergency medical assistance service ( SAMU), paramedical team and the emergency unit) will be included in the study. With the use of questionnaries, information will be collected from patients or witnesses by the SAMU, the paramedical team or physicians of the emergency unit. A 7-day follow-up will be carried out by the principal investigator (PI) of each center.

SUMMARY:
The occurrence of isolated or recurring epileptic seizures accounts for an important use of the healthcare system. Typically, epileptic patient will consult ten times a year a physician (specialist or familial doctor) and will justify 24 diagnostic procedures or additional examinations. Moreover, epileptic seizures are associated with frequent use of emergency departments. From the first emergency call received by the Emergency medical assistance service (SAMU), the actual management of the patient having epileptic seizure includes the eventual transfer to the paramedical team then within an emergency unit. However in some cases, emergency allocation may be avoided as 70% of patients recover their baseline condition upon admission. The main objective of this study is to describe the management of the adult population suffering from suspected seizure by the emergency structures. For 3 consecutive days, all patients with suspected epileptic seizures (diagnosed by the SAMU, paramedics and emergency unit) will be enrolled in the study. Data of medical care management and information from patients or witnesses will be collected on a questionnaire by the physicians of the SAMU, paramedics and emergency unit. Then, the anonymized questionnaires will be sent to RESUVAL (Emergency Network of the Rhone Valley) to ensure data entry and statistical analysis. By identifying the factors leading the SAMU to transfer a patient with suspected epileptic seizure to an emergency unit, this study will provide a more appropriate procedure to prevent unnecessary emergency admissions. It will also gain more insights into the patient outcomes, such as complementary medication, brain examination or referral to a neurologist.

DETAILED DESCRIPTION:
Epilepsy is a neurological disorder in which brain activity becomes abnormal, causing unpredictable seizures. It affects people of all ages and in 2018, it is estimated that 1% of the world's population is suffering from epilepsy. In France, the recommendations for care of people with a first or recurring seizures are now well codified (Société française de neurologie, 2014; Société française de Médecine d'Urgence, 2018). It is also recognized that the quality of the neurological follow-up and the subsequent control of epilepsy reduces the cost of medical care and the number of emergency entries (Manjunath, 2012). However, occurrence of epileptic seizures still accounts for an important use of the healthcare system and especially those of emergency unit. Typically, it has been reported that epileptic patient will consult ten times a year a physician (specialist or familial doctor) and will justify 24 diagnostic procedures or additional examinations (Kurth, 2010). In France, nearly 3% of calls to the Emergency medical assistance service (SAMU) and 1.6% of emergency entries are linked to an epileptic seizure. Moreover, the care and the management of epilepsy by the SAMU and emergency structures generate a significant financial cost. The French CAROLE cohort study described that in the first and second year after diagnosis of epilepsy, hospitalization cost respectively accounts for 68% and 40% of the total cost of care (de Zelicourt, 2000). In addition, it has been estimated that the extra cost of emergency admissions for patients with epilepsy represents $ 9.6 billion per year (Cramer, 2014). The decision of a physician to orient a patient toward an emergency unit is based on clinical or anamnesis criteria. An European study has highlighted factors associated with an increased risk of emergency admission (Balestrini, 2013); Patient with current psychiatric therapy, drug polytherapy, comorbidities, or that are experiencing more than one episode in the same day and changes in usual seizure pattern are more exposed to be referred to an emergency center (Balestrini, 2013). These findings were reinforced by another study showing the importance of ambulatory supervision measures in the prevention of emergency admissions not justified medically (Tatum, 2008). However, sociodemographic disparities in health care use among epileptic patients have been identified in the US, which could be explained by the executive differences of the sites of care (Begley, 2009). Such data on the practices in the emergency services nor the adequacy between practices and health recommendations are currently unavailable in France. However, we can assume that such heterogeneity of health care exists in France and leads to different health care management. Moreover, the significant emergency congestion that are collectively facing hospitals is associated with heterogeneity in patient health care (Wong, 2010). Although neuro-examination allows an adapted antiepileptic treatment when it is justified (Paliwal, 2015) and is required following episode of inaugural seizure, the possibility for a patient admitted in the emergency department to benefit from an electroencephalogram (EEG) has not been precisely studied in France. However, a study identified patterns (such as head trauma, neurovascular damage, infectious context, withdrawal context in antiepileptic drugs …) that lead to brain investigation by complementary neuroimaging (Annegers, 1995). Also, it has been reported that older patient have higher probability to benefit from neuroimaging (Martindale, 2011).

Finally, it is important to note that in some cases, emergency admissions may be avoided as 60% of patients have an already known historical diagnosis of epilepsy (Girot, 2015), 70% of patients recovered their baseline condition upon admission (Dickson, 2017) or other were discharged home without medical care (Dickson, 2017). In Australia, the prevalence of emergency presentations for recurring seizures has decreased and it is suggested to be linked with improved levels of education and health care delivery (Cordato, 2009).

Thus, we hypothesized that an optimized emergency medical pathway among epileptic patient would optimized the patient outcome (epilepsy treatments, quality of life) and would also benefit for the logistic of the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Any patient ≥18 years calling the SAMU and / or supported by a paramedical team and / or admitted to an emergency unit for suspected symptoms of epileptic seizure will be included.

  * SAMU=Emergency medical assistance service

Exclusion Criteria:

* Patients with no epileptic seizures (assessed by the SAMU, paramedical team and the emergency unit) can't be enrolled in the study.

  * SAMU=Emergency medical assistance service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient ≥18 years calling the Emergency medical assistance service (SAMU)
Sampling Method: Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Description of the management of the adult population suffering from suspected seizure by the emergency structures. | 3 days
  The patient journey will be followed from the call to the emergency medical assistance service (SAMU) with a possible transfer by the paramedical team until the care, within the emergency unit.

SECONDARY OUTCOMES:
The patient characteristics, treatment pathway and outcomes after discharge | 11 days
  The secondary objectives of the study will determine:
  * the factors leading the SAMU to transfer a patient with suspected epileptic seizure to an emergency unit.
  * the factors leading a paramedical physician or emergency physician to prescribe an emergency antiepileptic treatment and / or a complementary brain imaging (CT or MRI) examination,
  * if admission to the emergency department resulted in the immediate or delayed completion of an EEG or neurology consultation, and within what period of time,
  * the final diagnosis and its possible adequacy with the initial diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie MEYRAN, MD, Principal Investigator — Centre Hospitalier Saint Joseph St Luc de Lyon
Locations (1):
- Centre Hospitalier St Joseph St Luc, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided
The questionnaires contain personal data: age and sex of the patient, place of care, treatment and home address.